CLINICAL TRIAL: NCT01708213
Title: A Multi-center, Open-label, Prospective Study of Implanted Cross-linked HA Device, Aline HA, for Soft Tissue Augmentation, to Treat Only One Anatomic Feature in up to 100 Subjects for 6 Months
Brief Title: Safety Evaluation of Aline HA, an Implanted Cross-Linked HA Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TauTona Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 10664
Record Dates: First submitted 2012-10-12; First posted 2012-10-16 (Estimated); Results first posted 2014-12-17 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Disorder of Soft Tissue
Keywords: soft tissue; augmentation; correction; wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dermal Filler - Aline HA (Experimental): Single armed study
  Interventions: Device: Aline HA

INTERVENTIONS:
Device: Aline HA — Implantable dermal filler

SUMMARY:
The protocol hypothesis is that treatment with Aline HA™ will be safe through 6 months as determined by clinical assessment of treatment sites and routine tracking of adverse events.

DETAILED DESCRIPTION:
A multi-center, open-label, prospective study of implanted cross-linked HA device, Aline HA, for soft tissue augmentation, to treat only one anatomic feature in up to 100 subjects for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥ 21 and ≤ 70 years of age.
2. The patient must be willing and able to provide informed consent.
3. The patient must be able to read.
4. The patient is willing and able to comply with the study protocol.
5. The patient is seeking soft tissue augmentation
6. The patient has a pre-treatment Wrinkle Severity Score (WSS) ≥ 2 for any NLF to be treated.
7. The patient agrees to follow-up examinations out to 6 months post final treatment.

Exclusion Criteria:

* Exclusion Criteria: 1) The patient has had (or plans to have) cosmetic procedures to treat the intended treatment area, such as:

  1. Ablative or non-ablative resurfacing procedures including but not limited to medium depth or deeper chemical peeling, dermabrasion, laser resurfacing or fractional resurfacing that would affect the treatment area within the last 12 months.
  2. Laser or light based therapy that would affect the treatment area within the last 6 months.
  3. Face, neck or brow lift or other surgical procedure of the head and neck that would affect the treatment area in the last 18 months.
  4. Non-permanent dermal filler treatment in the treatment area within the last 9 months.
  5. Permanent implant or dermal filler treatment in the treatment area at any point in time.
  6. Neurotoxin treatment that would affect the treatment area in the last 6 months, if the treatment area is below the eyes.
  7. Neurotoxin treatment that would affect the treatment area in the last 9 months, if the treatment area is above the eyes.

     2) The patient has had or plans to use a pharmaceutical (topical or oral) anti-wrinkle product or other products (e.g., topical retinoids, hormone creams) affecting inflammation in the treatment area within 30 days of the study 3) The patient has inflammatory or infectious skin conditions or unhealed wounds in the treatment areas.

     4) The patient has a cancerous or pre-cancerous lesion and/or has had radiation exposure in the treatment area in the last 24 months.

     5) The patient has a history of anaphylaxis, multiple severe allergies, atopy, or is allergic to lidocaine or amide-based anesthetics, hyaluronic acid products, Streptococcal proteins or proteins from other gram positive organisms.

     6) The patient has a history of significant bleeding disorders. 7) The patient has scleroderma or fibrotic tissue disease. 8) The patient is female and of child bearing potential and/or is pregnant or lactating or is not using medically effective birth control, such as hormonal methods in use at least 30 days prior to implantation, or barrier methods such as a condom and spermicide in use at least 14 days prior to implantation.

     9) The patient is using a Legally Authorized Representative. 10) The patient is an employee or employee's family member of either the Study Sponsor or a Study Site.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2012-10; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nowell Solish, MD, Principal Investigator
Locations (2):
- Canada (2):
  - Dr. Nowell Solish, Toronto, Ontario
  - The Westmount Institute of Plastic Surgery, Montreal, Quebec

RESULTS

PARTICIPANT FLOW:
Groups:
- Dermal Filler - Aline HA: Non-Randomized
  Aline HA: Implantable dermal filler
Period: Overall Study
Arm/Group | Dermal Filler - Aline HA
Started | 72
Completed | 71
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Dermal Filler - Aline HA
Number analyzed (Participants) | 72
Age, Continuous [Mean (Full Range); unit: years] | 50.5 [34 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 8
Region of Enrollment [Number; unit: participants]
  Canada | 72

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Treatment Site Responses Post Procedure
Description: The primary endpoint of this study is to assess treatment site responses and adverse events through 6 months post procedure.
Time Frame: 6 months
Measure: Number; unit: percentage of participants with any AE
Arm/Group | Dermal Filler - Aline HA
Number analyzed (Participants) | 72
percentage of participants with any AE | 78

2. Secondary Outcome: Number of Participants With a Decrease in the Wrinkle Severity Scale for Nasolabial Folds
Description: For this study, a decrease (at least one point) in the rating, relative to pre-treatment rating, when assessed by Investigators at the 1-Month, 3-Month, and 6-Month visits was considered clinically significant (P value less than 0.05).
  WSS:
  (0) - No wrinkle
  1. - Just perceptible wrinkle
  2. - Shallow wrinkle
  3. - Moderately deep wrinkle
  4. - Deep wrinkle, well-defined edges
  5. - Very deep wrinkle, redundant fold
Time Frame: 6 months
Population: Wrinkle Severity Score (WSS) assessment values of the Nasolabial Folds treatment area for the Per Protocol population (N=10) is a subgroup of the N=43 per protocol subjects treated. Reporting on the subjects with a 1 point improvement on the WSS at 6 months time.
Measure: Number; unit: participants
Arm/Group | Dermal Filler - Aline HA
Number analyzed (Participants) | 10
participants | 5
Statistical Analysis 1: Comparison: Dermal Filler - Aline HA; Test type: Superiority or Other; p < 0.05, Parametric testing; Parametric Testing = 0.05

3. Secondary Outcome: Percentage of Participants That Were Satisfied With the Treatment as Rated by GAIS
Description: This was measured using the Global Aesthetic Improvement Scale (GAIS). With the Global Aesthetic Improvement Scale (GAIS Scale) results of 1, 2 and 3 at 6 months were considered satisfied in this study.
Time Frame: 6 months
Measure: Number; unit: percentage of participants
Arm/Group | Dermal Filler - Aline HA
Number analyzed (Participants) | 43
percentage of participants | 60

ADVERSE EVENTS:
Time Frame: 6 months
Description: As reported by the investigator or the subject
Groups:
- Dermal Filler - Aline HA: To evaluate the safety and performance of Aline HA to treat mild to severe wrinkles in adult subjects
Arm/Group | Dermal Filler - Aline HA
Serious Adverse Events (participants affected / at risk) | 0/72
Other Adverse Events (participants affected / at risk) | 56/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dermal Filler - Aline HA (N=72)
Administration Site Conditions (General disorders) | 53
Headache (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No